CLINICAL TRIAL: NCT00773500
Title: Impact of Vendor Systems on Ambulatory Medication Safety
Acronym: BWHCERT5E
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: U18HS0169705E
Record Dates: First submitted 2008-10-03; First posted 2008-10-16 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Medication Errors
Keywords: Medication Errors
MeSH Terms: interventions — Electronic Prescribing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Providers adopting electronic prescribing in New York City, New York
  Interventions: Other: Electronic prescribing
- 2: Providers adopting electronic prescribing in the Taconic region of New York
  Interventions: Other: Electronic prescribing

INTERVENTIONS:
Other: Electronic prescribing — Implementation of a commercially available electronic prescribing system with clinical decision support

SUMMARY:
Our objective is to determine the effects of electronic prescribing on medication safety including medication errors, near misses and preventable adverse drug events in the ambulatory setting. Study design will be a longitudinal evaluation of errors early after implementation and after sustained use.

DETAILED DESCRIPTION:
We will compare the effects of different vendor-based electronic prescribing systems on ambulatory medication safety in various settings, including rural and underserved areas and determine the effects of electronic prescribing systems on ambulatory medication safety over time.

ELIGIBILITY:
Inclusion Criteria:

* >=0.75 FTE providers

Exclusion Criteria:

* <0.75 FTE providers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study will take place in 2 NYS communities. We will select 2 communities in order to assemble a study population with the following characteristics: use of at least 2 different vendor-based systems, different implementation times (with some communities being early adopters and others experienced users), and inclusion of urban underserved and federally defined rural areas.
  We will select the following 2 communities/organizations: the community health centers implementing electronic prescribing with the New York City Department of Health (NYC DOH) and the Taconic Health Information Network and Community (THINC) in the Hudson Valley of New York. Both communities have expressed their interest in participating in this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
prescribing error | 1 year

SECONDARY OUTCOMES:
near misses | 1 year
preventable adverse drug events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rainu Kaushal, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Taconic IPA, Fishkill, New York
  - New York City Department of Health and Mental Hygiene, New York, New York

REFERENCES:
- [Derived] Abramson EL, Pfoh ER, Barron Y, Quaresimo J, Kaushal R. The effects of electronic prescribing by community-based providers on ambulatory medication safety. Jt Comm J Qual Patient Saf. 2013 Dec;39(12):545-52. doi: 10.1016/s1553-7250(13)39070-9. PMID 24416945